CLINICAL TRIAL: NCT03803618
Title: Effectiveness of the Tetravalent Dengue Vaccine, CYD-TDV (Dengvaxia®) in the Philippines
Brief Title: Dengue Effectiveness Study in the Philippines
Status: Completed | Type: Observational
Sponsor: University of the Philippines (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry); Research Institute for Tropical Medicine, Philippines (Other Government)
Responsible Party: Sponsor
Other Study IDs: UPM REB 2017-0237
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Dengue; Severe Dengue; Virologically Confirmed Dengue
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Any leftover sera will be used for future studies and stored at UPM-NIH for fifteen (15) years after the end of this study. Future studies using the sera will undergo appropriate ethical reviews as required. After this period, specimens will be destroyed according to local guidelines. Additional consent will be obtained from the parent for storage and future use of these samples. Only the Principal Investigator and designated study personnel will have access to these specimens.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Confirmed dengue case: Dengue cases who are 9-14 years old during the dengue mass vaccination program in Cebu with <5 days history of fever, admitted in the participating hospitals with dengue virus confirmation by RT-PCR
- Control: Age and sex matched neighborhood controls

SUMMARY:
This is an observational study that aims to determine the effectiveness of a tetravalent dengue vaccine (CYD-TDV) when given through a community-based immunization program against hospitalized and /or severe virologically confirmed dengue.

DETAILED DESCRIPTION:
This is a matched case-control study. Cases will be children who are admitted with a clinical suspicion of dengue at the study hospitals and were eligible to have received the dengue vaccine during the mass immunization. The outcome of interest is hospitalized and/or severe virologically-confirmed dengue and the exposure is receipt of the dengue vaccine. Each case will be matched to two controls who were also eligible to have received the dengue vaccine and lives in the same area as the case. Cases and controls will be matched by age and sex.

ELIGIBILITY:
Inclusion Criteria:

CASE-CONTROL STUDIES

* For a suspected case to be enrolled in the study, he/she should:

  * Provide signed informed consent and assent (as applicable)
  * Be within the age group eligible to receive the dengue vaccine at the time of mass vaccination (i.e. no condition that would have made him/her ineligible for dengue vaccination)
  * Be admitted in any of the participating hospitals for suspected dengue
  * Have ≤5 days history of fever.
  * For the case to be included in the analysis, the participant must meet all the inclusion criteria above plus have virologically-confirmed dengue infection by RT-PCR
* For controls to be recruited into the study, he/she should:

  * Provide signed informed consent and assent (as applicable)
  * Be age and sex-matched to the case
  * Be from the same community as the matched case
  * Be eligible to have received dengue vaccine during the community-based dengue immunization campaign in 2017 (i.e. no condition that would have made him/her ineligible for dengue vaccination)
  * Have had no episode of clinically-diagnosed or laboratory-confirmed dengue fever from the start of the community -based dengue immunization campaign to the focal time (the date of onset of dengue fever in the matched case)
  * Should not have been previously recruited as a control.

Exclusion Criteria:

• Any subject whose parent/guardian refuse to provide informed consent and/or assent.

* In addition, the following conditions automatically exclude children from the dengue mass immunization:

  * Children <9 years or adults older than 45 years of age
  * Anyone who is allergic or has had an allergic reaction to a prior dose or to any component of the dengue vaccine
  * Recipient of blood product in the last 3 months
  * Immunocompromised individuals, due to but not limited to genetic defects, HIV infection, or therapies that affect the immune system such as high-dose corticosteroids or chemotherapy
  * Recipient of any vaccine within the past month
  * History of bleeding disorder
  * Pregnant or breastfeeding women
  * Enrolled in dengue vaccine Phase 3 clinical study

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Individuals to be enrolled in the study as probable cases will be admitted patients in the hospital study sites who are residents of the area, eligible to have received the dengue vaccine at the time of the initiation of community-based dengue vaccination program, and suspected to have dengue.
Sampling Method: Non-Probability Sample
Enrollment: 2081 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
hospitalized and / or severe virologically confirmed dengue | 5 years
  The primary outcome are children who are hospitalized and/or severe virologically confirmed dengue

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline L. Deen, MD, Principal Investigator — UPM - NIH, Institute of Child Health and Human Development
Locations (4):
- Philippines (4):
  - Cebu Provincial Hospital - Balamban, Balamban, Cebu
  - Cebu Provincial Hospital - Bogo, Bogo, Cebu
  - Cebu Provincial Hospital - Danao, Danao, Cebu
  - Eversley Childs Sanitarium and General Hospital, Mandaue City, Cebu